CLINICAL TRIAL: NCT06644794
Title: Comparison of Progesterone-modified Natural Cycle and Hormone Replacement Therapy Cycle for Endometrial Preparation in Single Frozen Blastocyst Transfer
Brief Title: Progesterone-modified Natural Cycle for FET
Acronym: COMPROSET
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jing-Yan Song, Prof., Shandong University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P4mNC@SDUTCM
Record Dates: First submitted 2024-10-12; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Infertility, Female
Keywords: Progesterone-modified natural cycle; Hormone replacement therapy; Frozen-thawed embryo transfer
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P4mNC group (Experimental): On days 8-12 of the menstrual cycle (MC), depending on the length of the patient's MC, transvaginal ultrasound is used to monitor follicular development and endometrial growth. Vaginal micronized progesterone (Utrogestan, Besins, Belgium) is started at 200 mg in the afternoon and 200 mg in the evening when the dominant follicle reached ≥16 mm and the endometrial thickness is at least 7 mm. A blastocyst is transferred on day 5 after the addition of progesterone. On day 14 after blastocyst transfer, serum β-hCG levels are measured. Upon positive serum pregnancy testing, progesterone support will continue until 8-10 weeks of gestation. However, afternoon progesterone use is eliminated for 30 days after embryo transfer.
  Interventions: Drug: Progesterone-modified natural cycle preparation for frozen embryo transfer
- HRT group (Active Comparator): Endometrial preparation will begin on the second day of the menstrual cycle with oral estradiol (E2) valerate at a dose of 2 mg twice daily. When the patient's endometrial thickness is ≥7 mm, vaginal progesterone administration will be initiated at a dose of 200 mg 3 times daily. On day 5 of the progesterone administration, blastocysts are thawed and transferred. For patients with endometrial thickness <7 mm, patients continued oral E2 until the endometrium is ≥7 mm. On day 14 after blastocyst transfer, serum β-hCG levels are measured. Upon positive serum pregnancy testing, E2 and progesterone supplementation is continued for 8-10 weeks of gestation.
  Interventions: Drug: Hormone replacement therapy cycle preparation for frozen embryo transfer

INTERVENTIONS:
Drug: Progesterone-modified natural cycle preparation for frozen embryo transfer — A novel endometrial preparation protocol that optimizes the natural cycle, whereby as long as the thickness of the endometrium is suitable for embryo transfer, vaginal progesterone can be used to transform the endometrium before ovulation and subsequently FET.
  Arms: P4mNC group
Drug: Hormone replacement therapy cycle preparation for frozen embryo transfer — A traditional endometrial preparation protocol is used for FET, which involves using fixed or flexible exogenous estradiol for artificial cycles. This protocol typically involves starting exogenous estradiol on day 3 or 4 of the cycle, continuing for 7-10 days, and then discontinuing. Upon determining that the endometrial thickness meets the standard, progesterone conversion of the endometrium can be performed.
  Arms: HRT group

SUMMARY:
Hormone replacement therapy (HRT) cycles, despite the ease of synchronizing embryo thawing and embryo transfer timing, increase the risk of pregnancies and obstetric complications compared to natural cycles (NC). By ensuring the presence of the corpus luteum while reducing the number of monitoring sessions, the progesterone modified natural cycle (P4mNC) offers more convenience for the patient than the normal NC. This study is designed to compare the effects of P4mNC and HRT cycles on FET outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 to 44 years undergoing FBT
* Body mass index (BMI) 18-35 kg/m2
* Having regular ovulatory cycles

Exclusion Criteria:

* Untreated uterine adhesions
* Medical contraindications to estrogen and progesterone therapy
* Illnesses contraindicating assisted reproductive technology or pregnancy
* History of recurrent implantation failures (> 2 embryo transfer failures)

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Live birth | Within 1 year after randomization
  A live birth is defined as the delivery of any surviving newborn at 28 weeks or more of gestation.

SECONDARY OUTCOMES:
Biochemical pregnancy | Two weeks after embryo transfer
  Serum level of ß-hCG > 50 mIU/mL
Clinical pregnancy | Five weeks after embryo transfer
  Fetal heartbeat observed by vaginal ultrasound
Ongoing pregnancy | Ten weeks after embryo transfer
  The presence of a gestational sac and fetal heartbeat after 12 weeks of gestation
Miscarriage | Within 28 weeks of pregnancy
  A condition in which the embryo or fetus does not survive and is not spontaneously absorbed or expelled from the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Gao Sun, MD, Principal Investigator — Shandong University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Inhorn MC, Patrizio P. Infertility around the globe: new thinking on gender, reproductive technologies and global movements in the 21st century. Hum Reprod Update. 2015 Jul-Aug;21(4):411-26. doi: 10.1093/humupd/dmv016. Epub 2015 Mar 22. PMID 25801630
- [Background] Mascarenhas MN, Cheung H, Mathers CD, Stevens GA. Measuring infertility in populations: constructing a standard definition for use with demographic and reproductive health surveys. Popul Health Metr. 2012 Aug 31;10(1):17. doi: 10.1186/1478-7954-10-17. PMID 22938182
- [Background] Doody KJ. Cryopreservation and delayed embryo transfer-assisted reproductive technology registry and reporting implications. Fertil Steril. 2014 Jul;102(1):27-31. doi: 10.1016/j.fertnstert.2014.04.048. Epub 2014 Jun 4. PMID 24907917
- [Background] Zhang Y, Fu X, Gao S, Gao S, Gao S, Ma J, Chen ZJ. Preparation of the endometrium for frozen embryo transfer: an update on clinical practices. Reprod Biol Endocrinol. 2023 Jun 8;21(1):52. doi: 10.1186/s12958-023-01106-5. PMID 37291605
- [Background] Roelens C, Blockeel C. Impact of different endometrial preparation protocols before frozen embryo transfer on pregnancy outcomes: a review. Fertil Steril. 2022 Nov;118(5):820-827. doi: 10.1016/j.fertnstert.2022.09.003. PMID 36273850
- [Background] Gu F, Wu Y, Tan M, Hu R, Chen Y, Li X, Lin B, Duan Y, Zhou C, Li P, Ma W, Xu Y. Programmed frozen embryo transfer cycle increased risk of hypertensive disorders of pregnancy: a multicenter cohort study in ovulatory women. Am J Obstet Gynecol MFM. 2023 Jan;5(1):100752. doi: 10.1016/j.ajogmf.2022.100752. Epub 2022 Sep 15. PMID 36115572
- [Background] von Versen-Hoynck F, Schaub AM, Chi YY, Chiu KH, Liu J, Lingis M, Stan Williams R, Rhoton-Vlasak A, Nichols WW, Fleischmann RR, Zhang W, Winn VD, Segal MS, Conrad KP, Baker VL. Increased Preeclampsia Risk and Reduced Aortic Compliance With In Vitro Fertilization Cycles in the Absence of a Corpus Luteum. Hypertension. 2019 Mar;73(3):640-649. doi: 10.1161/HYPERTENSIONAHA.118.12043. PMID 30636552
- [Background] Kornilov N, Polyakov A, Mungalova A, Yakovleva L, Yakovlev P. Progesterone-modified natural cycle preparation for frozen embryo transfer. Reprod Biomed Online. 2024 Nov;49(5):104350. doi: 10.1016/j.rbmo.2024.104350. Epub 2024 Jul 2. PMID 39244908
- [Derived] Yuan HN, Song JY, Sun ZG. Comparison of progesterone-modified natural cycle and hormone replacement therapy cycle for endometrial preparation in single frozen blastocyst transfer (COMPROSET): protocol for an open-label randomized controlled trial. Front Med (Lausanne). 2025 Apr 28;12:1522004. doi: 10.3389/fmed.2025.1522004. eCollection 2025. PMID 40357273